CLINICAL TRIAL: NCT05836051
Title: Testing the Effect of ENDS Flavors on Neurotransmission
Acronym: TEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andrea Hobkirk, PhD, Assistant Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 19883; 24844; R61DA056764 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Dependence
Keywords: Tobacco; Nicotine; Smoking; Addiction
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Behavior, Addictive | interventions — Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hexyl Acetate (Experimental): E-cigarette liquid containing hexyl acetate, ethyl maltol, propylene glycol, vegetable glycerin and methylbutyl acetate with nicotine salt.
  Interventions: Other: Flavor
- Ethyl Acetate (Active Comparator): E-cigarette liquid containing ethyl acetate, ethyl maltol, propylene glycol, vegetable glycerin and methylbutyl acetate with nicotine salt.
  Interventions: Other: Flavor

INTERVENTIONS:
Other: Flavor — E-liquid flavor chemicals

SUMMARY:
The overarching goal of this translational proposal is to determine if neuroactive flavor chemicals can enhance the addiction potential of electronic nicotine delivery systems (ENDS) by altering brain function and behavior.

DETAILED DESCRIPTION:
For this randomized double-blind controlled trial, tobacco users will be randomized to use ENDS with an e-liquid containing a neuroactive flavor (hexyl acetate) vs. an inactive flavor (ethyl acetate) for ten days as a supplement to their typical tobacco use. Laboratory measures of ENDS reinforcement, subjective ENDS ratings, and brain reactivity to the flavor using functional magnetic resonance imaging (fMRI) will be collected at baseline and after ten days of ENDS use.

ELIGIBILITY:
Inclusion Criteria:

1. 21 to 60 years old
2. Regular users of inhaled tobacco products (≥5 days out of the last 28)
3. Not planning to quit tobacco use within next month
4. Able to read and write in English

Exclusion Criteria:

1. Major neurological conditions or brain trauma
2. Current substance use impairing participation
3. Unstable or significant medical conditions (e.g., COPD, coronary heart disease)
4. Current use of smoking cessation medication (e.g., varenicline, patch)
5. Uncontrolled serious mental illness, suicidality, or inpatient psychiatric hospitalization in the past 6 months
6. Known allergic reaction to ENDS liquids ingredients propylene glycol or vegetable glycerin
7. Unable to use study provided ENDS ad-libitum for at least 3 hours per day
8. Pregnant or breastfeeding as indicated by self-report or urine pregnancy screen

MRI-specific exclusion criteria:

1. MRI safety contraindications (e.g., metal implants, claustrophobia)
2. Major neurological conditions or brain trauma

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Brain reward reactivity | Pre to post-intervention (approximately 10 days)
  Brain reward reactivity will be calculated as the percent change in average blood oxygen-level dependent (BOLD) signal in a pre-defined ventral tegmental area (VTA) region of interest during ENDS inhalation
Absolute reinforcement | Pre to post-intervention (approximately 10 days)
  Absolute reinforcement will be calculated as the change in the average number of puffs per day during a 10-day use period

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not have explicit plans to share IPD on open-access or publicly accessible repositories. However, IPD will be de-identified and formatted along with codebooks to facilitate data sharing with investigators upon request and after the completion of a Data Use Agreement.